CLINICAL TRIAL: NCT01217814
Title: A Randomized, Double-blind, Parallel-group, Placebo- and Active Calibrator-controlled Study Assessing the Clinical Benefit of SAR153191 Subcutaneous (SC) on Top of MTX in Patients With Active RA Who Have Failed Previous TNF-α Antagonists
Brief Title: Effect of SAR153191 (REGN88) With Methotrexate in Patients With Active Rheumatoid Arthritis Who Failed TNF-α Blockers
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Due to delay in the study and the impact on the development timelines, not due to any identified safety concerns
Sponsor: Sanofi (Industry)
Collaborators: Regeneron Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: ACT11575; 2010-021020-94 (EudraCT Number); U1111-1115-3763 (Other: UTN)
Record Dates: First submitted 2010-10-07; First posted 2010-10-08 (Estimated); Results first posted 2017-09-01 (Actual); Last update posted 2017-09-01 (Actual); Status verified 2017-07

CONDITIONS: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — sarilumab; golimumab; Methotrexate; Leucovorin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Placebo (Placebo Comparator): Placebo 2 mL to match sarilumab once a week (qw) and 0.5 mL to match golimumab every 4 weeks (q4w) on top of MTX (15-25 mg) qw for 12 weeks.
  Interventions: Drug: Placebo; Drug: methotrexate (MTX); Drug: Folic/folinic acid
- Golimumab 50 mg (Active Comparator): Golimumab 50 mg q4w and placebo (matched to sarilumab) qw on top of MTX (15-25 mg) qw for 12 weeks.
  Interventions: Drug: Placebo; Drug: Golimumab; Drug: methotrexate (MTX); Drug: Folic/folinic acid
- Sarilumab 150 mg (Experimental): Sarilumab 150 mg qw and placebo (matched to golimumab) q4w on top of MTX (15-25 mg) qw for 12 weeks.
  Interventions: Drug: Sarilumab; Drug: Placebo; Drug: methotrexate (MTX); Drug: Folic/folinic acid

INTERVENTIONS:
Drug: Sarilumab — Pharmaceutical form: solution for injection
  Route of administration: subcutaneous
  Other Names: SAR153191; REGN88
  Arms: Sarilumab 150 mg
Drug: Placebo — Pharmaceutical form: solution for injection
  Route of administration: subcutaneous
Drug: Golimumab — Pharmaceutical form: solution for injection
  Route of administration: subcutaneous
  Other Names: Simponi®
  Arms: Golimumab 50 mg
Drug: methotrexate (MTX) — Pharmaceutical form: tablet or solution for injection
  Route of administration: Oral (tablet) or subcutaneous, intramuscular (solution)
Drug: Folic/folinic acid — Pharmaceutical form: tablet
  Route of administration: oral Folic/folinic acid continued according to local standard.

SUMMARY:
Primary Objective:

- To demonstrate that sarilumab (SAR153191/REGN88) on top of methotrexate (MTX) was superior in efficacy to placebo for the relief of signs and symptoms of rheumatoid arthritis (RA), in participants with active RA who had failed up to 2 tumor necrosis factor-alpha (TNF-α) antagonists.

Secondary Objectives:

* To assess the safety of sarilumab;
* To document the pharmacokinetic profile of sarilumab.

DETAILED DESCRIPTION:
The duration of the study period for each participant was approximately 22 weeks; including up to 4 weeks screening period, 12-week double-blind treatment period and 6-week safety follow-up period.

Participants who completed the 12-week treatment period were offered enrollment in a separate long-term extension study (LTS11210/NCT01146652).

ELIGIBILITY:
Inclusion criteria:

* Diagnosis of rheumatoid arthritis ≥6 months duration and American College of Rheumatology (ACR) Class I-III functional status at screening and baseline visits;
* Active disease defined as:

  * At least 6 of 68 tender joints and 6 of 66 swollen joints at screening and baseline visits, and
  * hs-C-Reactive Protein (hs-CRP) >10 g/L or Erythrocyte Sedimentation Rate (ESR) >28 mm/hr at screening visit;
* Continuous treatment with Methotrexate for at least 12 weeks and on stable dose (minimum 10 mg/week) for at least 6 weeks prior to the screening visit;
* Participant considered as Primary TNF-α blocker nonresponder. i.e.:

  * Appropriate for previous TNF-α blocker therapy
  * Lack of adequate clinical response after at least 3 months TNF-α blocker therapy with MTX or other synthetic disease modifying anti-rheumatic drug (DMARD) co-therapy.

Exclusion criteria:

* Age <18 years or >75 years;
* Pregnant or breastfeeding woman or woman of childbearing potential, unwilling to utilize adequate contraception or not to become pregnant during the entire study;
* Fever (>38°C), or chronic, persistent, or recurring infection(s);
* History of demyelinating disease;
* Current underlying hepatobiliary disease.

The above information was not intended to contain all considerations relevant to a participant's potential participation in a clinical trial.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2010-11; Primary Completion 2011-09 (Actual); Study Completion 2011-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi
Locations (14):
- United States (4):
  - Investigational Site Number 840026, Freehold, New Jersey
  - Investigational Site Number 840043, New York, New York
  - Investigational Site Number 840025, Jackson, Tennessee
  - Investigational Site Number 840038, Austin, Texas
- Colombia (3):
  - Investigational Site Number 170004, Barranquilla
  - Investigational Site Number 170005, Barranquilla
  - Investigational Site Number 170007, Bucaramanga
- Investigational Site Number 203002, Uherské Hradiště, Czechia
- Italy (2):
  - Investigational Site Number 380002, Florence
  - Investigational Site Number 380005, Genova
- Mexico (2):
  - Investigational Site Number 484008, Durango
  - Investigational Site Number 484002, Guadalajara
- Spain (2):
  - Investigational Site Number 724004, Oviedo
  - Investigational Site Number 724002, Valencia

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at 10 centers in United States and Europe. A total of 41 participants were screened between 15 November 2010 and 18 May 2011 of whom 16 participants were randomized and 25 were screen failures. Screen failures were mainly due to exclusion criteria met.
Pre-assignment Details: Participants were randomized 2:1:2 (Sarilumab 150 mg : Placebo : Golimumab 50 mg) via a centralized randomization system using an interactive voice response system stratified by region and number of previous anti-tumor necrosis factor-alpha (TNF-α) therapy.
Groups:
- Placebo: Subcutaneous (SC) injection of placebo 2 mL once a week (qw) to match sarilumab and 0.5 mL every 4 weeks (q4w) to match golimumab on top of methotrexate (MTX) (15-25 mg) qw for 12 weeks.
- Golimumab 50 mg: Golimumab 50 mg SC injection q4w and placebo (matched to sarilumab) SC injection qw on top of MTX (15-25 mg) qw for 12 weeks.
- Sarilumab 150 mg: Sarilumab 150 mg SC injection qw and placebo (matched to golimumab) SC injection q4w on top of MTX (15-25 mg) qw for 12 weeks.
Period: Overall Study
Arm/Group | Placebo | Golimumab 50 mg | Sarilumab 150 mg
Started | 4 | 5 | 7
Completed | 3 | 4 | 6
Not Completed | 1 | 1 | 1
Not completed — Adverse Event | 1 | 1 | 0
Not completed — Lack of Efficacy | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Placebo: SC injection of placebo 2 mL qw to match sarilumab and 0.5 mL q4w to match golimumab on top of MTX (15-25 mg) qw for 12 weeks.
- Total: Total of all reporting groups
Arm/Group | Placebo | Golimumab 50 mg | Sarilumab 150 mg | Total
Number analyzed (Participants) | 4 | 5 | 7 | 16
Age, Continuous [Mean (Standard Deviation); unit: years] | 45.3 (17.9) | 62.6 (7.6) | 54.0 (11.1) | 54.5 (13.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 3 | 7 | 14
  Male | 0 | 2 | 0 | 2

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Who Achieved at Least 20% Improvement in American College of Rheumatology (ACR20) Core Set Disease Activity Index at Week 12
Time Frame: Week 12
Population: As the number of participants randomized fell well below target (16 vs. 250), the efficacy data were not systematically collected or cleaned and no datasets have been created to report.
Arm/Group | Placebo | Golimumab 50 mg | Sarilumab 150 mg
Number analyzed (Participants) | 0 | 0 | 0

2. Secondary Outcome: Percentage of Participants Who Achieved at Least 50% Improvement in American College of Rheumatology (ACR50) Core Set Disease Activity Index at Week 12
Time Frame: Week 12
Population: as for outcome 1
Arm/Group | Placebo | Golimumab 50 mg | Sarilumab 150 mg
Number analyzed (Participants) | 0 | 0 | 0

3. Secondary Outcome: Percentage of Participants Who Achieved at Least 70% Improvement in American College of Rheumatology Core (ACR70) Set Disease Activity Index at Week 12
Time Frame: Week 12
Population: as for outcome 1
Arm/Group | Placebo | Golimumab 50 mg | Sarilumab 150 mg
Number analyzed (Participants) | 0 | 0 | 0

4. Secondary Outcome: Disease Activity Score for 28 Joints (DAS28) at Week 12
Time Frame: Week 12
Population: as for outcome 1
Arm/Group | Placebo | Golimumab 50 mg | Sarilumab 150 mg
Number analyzed (Participants) | 0 | 0 | 0

5. Secondary Outcome: European League Against Rheumatism (EULAR) Response at Week 12
Time Frame: Week 12
Population: as for outcome 1
Arm/Group | Placebo | Golimumab 50 mg | Sarilumab 150 mg
Number analyzed (Participants) | 0 | 0 | 0

6. Secondary Outcome: Percentage of Participants Achieving DAS28 Remission Score < 2.6 at Week 12
Time Frame: Week 12
Population: as for outcome 1
Arm/Group | Placebo | Golimumab 50 mg | Sarilumab 150 mg
Number analyzed (Participants) | 0 | 0 | 0

7. Secondary Outcome: Pharmacokinetic (PK) Parameter: Serum Concentration of Functional and Bound Sarilumab
Time Frame: Week 12
Population: Analysis was performed in PK population of all participants with at least one non-missing serum concentration data.
Measure: Mean (Standard Deviation); unit: ng/mL
Groups:
- Sarilumab 150 mg qw: Sarilumab 150 mg SC injection qw and placebo (matched to golimumab) SC injection q4w on top of MTX (15-25 mg) qw for 12 weeks.
Arm/Group | Sarilumab 150 mg qw
Number analyzed (Participants) | 7
ng/mL
  Bound Concentration | 4271.43 (1328.86)
  Functional Concentration | 42391.43 (26168.68)

ADVERSE EVENTS:
Time Frame: All Adverse Events (AE) were collected from signature of the informed consent form up to the final visit (week 18) regardless of seriousness or relationship to investigational product.
Description: Reported adverse events are treatment-emergent adverse events that is AEs that developed/worsened during the 'on treatment period' (time from the first dose injection of the double-blind investigational product to the end of the follow-up period).
Arm/Group | Placebo | Golimumab 50 mg | Sarilumab 150 mg
Serious Adverse Events (participants affected / at risk) | 0/4 | 0/5 | 0/7
Other Adverse Events (participants affected / at risk) | 3/4 | 1/5 | 3/7
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=4) | Golimumab 50 mg (N=5) | Sarilumab 150 mg (N=7)
Influenza (Infections and infestations) | 0 | 0 | 1
Nasopharyngitis (Infections and infestations) | 1 | 0 | 0
Sinusitis (Infections and infestations) | 1 | 0 | 0
Urinary tract infection (Infections and infestations) | 1 | 0 | 0
Hypertension (Vascular disorders) | 0 | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 0 | 1 | 0
Vomiting (Gastrointestinal disorders) | 0 | 1 | 0
Dermatitis (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Application site reaction (General disorders) | 0 | 0 | 1
Chills (General disorders) | 0 | 0 | 1
Transaminases increased (Investigations) | 0 | 0 | 1
Accidental overdose (Injury, poisoning and procedural complications) | 1 | 0 | 1

LIMITATIONS AND CAVEATS:
The study was prematurely terminated due to small number of participants entering randomization.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If no publication has occurred within 12 months of the completion of the study, the Investigator shall have the right to publish/present independently the results of the study. The Investigator shall provide the Sponsor with a copy of any such presentation/publication for comment at least 30 days before any presentation/submission for publication. If requested by the Sponsor, any presentation/submission shall be delayed up to 90 days, to allow the Sponsor to preserve its proprietary rights.